CLINICAL TRIAL: NCT02543047
Title: THE ANGIOSHIELD STUDY:Feasibility Study to Demonstrate the Safety of the Angioshield System to Provide Mechanical Support for Vein Grafts Used in CABG Surgery
Brief Title: The Angioshield Study Feasibility II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neograft Technologies, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP14-026
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right Region (Active Comparator): Angioshield will be applied to provide Mechanical Support for Vein Grafts Used in CABG in the right region of the heart
  Interventions: Device: Angioshield
- Left Region (Active Comparator): Angioshield will be applied to provide Mechanical Support for Vein Grafts Used in CABG in the left region of the heart
  Interventions: Device: Angioshield

INTERVENTIONS:
Device: Angioshield — Angioshield is applied to vein graft to provide Mechanical Support for Vein Grafts Used in CABG Surgery

SUMMARY:
Feasibility Study to Demonstrate the Safety of the Angioshield System to Provide Mechanical Support for Vein Grafts Used in CABG Surgery.

DETAILED DESCRIPTION:
The study is designed to investigate the feasibility of using an applied support (Angioshield) to a saphenous vein to be used in Coronary Artery Bypass Surgery. It is a feasibility to determine safety prior to launching a larger pivotal study. The primary endpoint, 30-day safety, will be assessed by recording and reporting of adverse events during surgery and throughout the investigation until the 30-day follow-up visit. The secondary endpoints, long term safety and patency, will be assessed by recording and reporting of adverse events and graft patency (via serial CT angiograms) at the 30, 90, and 365 day follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

Subject will be eligible for inclusion in the investigation if he/she:

1. is between the ages of 18 and 80 years of age, inclusive
2. requires CABG surgery due to atherosclerotic coronary artery disease with minimum of two SVGs, one used to bypass a stenosis in the main Right Coronary artery and one used to bypass a stenosis in the Circumflex artery territory
3. is able to give their informed written consent
4. is willing and able to complete all follow-up visits and procedures
5. is to be treated via a medial sternotomy with cardio-pulmonary bypass during surgery
6. has adequate saphenous veins
7. Is a candidate for transcatheter therapy, PCI

Exclusion Criteria:

Subject will be excluded from participation in the investigation if he/she:

1. is currently enrolled in another clinical investigation
2. is unable to tolerate or comply with required post-surgical medications or imaging (e.g., anticoagulation regimen; or known allergy to contrast agent)
3. is or may be pregnant or is lactating, or plans to become pregnant in the next 12 months
4. history of a hypercoagulable state
5. has had an acute MI within the last 21 days
6. has had a previous CABG
7. requires emergency surgery
8. has a left ventricular ejection fraction (LVEF) less than 35 %
9. has a target vessel stenosis of less than 75%
10. has a transmural infarct of the target artery territory
11. has a serum creatinine greater than 1.5 mg/dL
12. is having concomitant -surgery of any kind
13. has had previous saphenectomy (See inclusion)
14. has saphenous vein sizes incompatible with treatment range (i.e., <3.5 mm or >5 mm inner diameter)
15. limb Ischemia or non-healing ulcer
16. has moderate to severe COPD defined as FEV 1 of less than 1 liter
17. has had a CVA in last 90 days
18. has diffuse disease in target vessel with an inadequate anastomotic touchdown site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Safety-reported MACE | 30 days
  The primary endpoint, 30 day safety, (MACE) will be assessed by recording and reporting of adverse events during surgery and throughout the investigation until the 30-day follow-up visit

SECONDARY OUTCOMES:
Safety, (MACE) will be assessed by recording and reporting of adverse events at the 30, 90, and 365 day follow-up visits. | 90 and 365 days
Patency: Graft patency (via serial CT angiograms) will be measured at the 30, 90, and 365 day follow-up visits. | 30, 90 ,and 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Gintaras Kalinauskas, MD, Principal Investigator — Santariskiu University Hospital
Locations (1):
- Santariskiu University Hospital, Vilnius, Lithuania